CLINICAL TRIAL: NCT05281250
Title: Evaluation of Physical Exercise as a Protective Factor for the Loss of Functional Capacity in Patients With Metastatic Tumors During Hospitalization. Pilot Study (EFFAPRO)
Brief Title: Evaluation of Physical Exercise to Prevent Functional Deterioration During Hospitalization (EFFAPRO)
Acronym: EFFAPRO
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: structural change at the hospital
Sponsor: Puerta de Hierro University Hospital (Other)
Responsible Party: Principal Investigator, Ana Ruiz-Casado, Medical Oncologist, Puerta de Hierro University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PH-07
Record Dates: First submitted 2018-08-27; First posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Cancer Patients; Hospitalized
Keywords: rehabilitation; physical activity; Physical condition
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised physical exercise (Experimental): Supervised exercise (aerobic + strength + flexibility) depending on the functional capacity of each patient, during hospitalization
  Interventions: Other: Supervised physical exercise
- Control (No Intervention): Patients will receive recommendations about exercising during hospitalization.

INTERVENTIONS:
Other: Supervised physical exercise — A supervised exercise is randomized. Although this intervention is not standard in our setting, it is a recommended practice, since it is known that rehabilitation strategies in hospitalized patients have different benefits.
  Arms: Supervised physical exercise

SUMMARY:
This is a randomized study that will measure the possible benefit of supervised training during the hospitalization of patients with stage IV neoplasms in active treatment.

DETAILED DESCRIPTION:
The trial is not going to be runned

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage IV neoplasms.
* Active treatment: chemotherapy, hormone therapy, immunotherapy or targeted therapies.
* Hospitalization at Medical Oncology Departmentof the Hospital Puerta de Hierro.
* Reason for hospitalization is expected to be solved in less than two weeks.

Exclusion Criteria:

* Patients who do not wish to participate.
* Cognitive impairment.
* Hospitalization due to progression of oncological disease.
* Acute coronary syndrome or bone fracture in limbs during the previous three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2018-08-28 (Actual); Study Completion 2018-08-28 (Actual)

PRIMARY OUTCOMES:
Functional capacity | Through study completion (average 10 days)
  Functional Independence Measure (FIM)

SECONDARY OUTCOMES:
Strength | Through study completion (average 10 days).
  Dynamometry
Cardiorespiratory condition | Through study completion (average 10 days)
  Six minute test .
Daily physical activity | Through study completion (average 10 days)
  Accelerometry during the hospitalization.
Fatigue-FACIT | Through study completion (average 10 days)
  FACIT Fatigue Scale
Fatigue-PERFORM | Through study completion (average 10 days)
  PERFORM Fatigue questionnaire (12-60) Higher, better (less fatigue)
Life quality: Q30 questionnaire | Through study completion (average 10 days)
  QLQ30 questionnaire (quality of life). 0-100 (HIGHER, better)
Anxiety and depression | Through study completion (average 10 days)
  HADS questionnaire (anxiety and depression). 0-42 (less better)
Length of hospital stay | Through study completion (average 10 days).
  Number of days the patient is hospitalized.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Ruiz Casado, Principal Investigator — Puerta de Hierro University Hospital
Locations (1):
- Hospital Universitario Puerta de Hierro, Majadahonda, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No